CLINICAL TRIAL: NCT06876662
Title: Long-Term Safety of Pirtobrutinib in Participants From Study LOXO-BTK-18001 With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma or Non-Hodgkin Lymphoma
Brief Title: A Study of (LY3527727) Pirtobrutinib in Participants With Previously Treated Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma or Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27289; 2024-517760-29-00 (EU CTIS Number); J2N-MC-JZ01 (Other: Eli Lilly and Company); J2N-MC-JZNY (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — pirtobrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JZ01 Pirtobrutinib (Experimental): Participants receive pirtobrutinib as defined in the originator study (LOXO-BTK-18001/J2N-OX-JZNA).
  Pirtobrutinib administered orally.
  Interventions: Drug: Pirtobrutinib

INTERVENTIONS:
Drug: Pirtobrutinib — Administered orally.
  Other Names: LOXO-305; LY3527727

SUMMARY:
Study J2N-MC-JZ01 (JZ01) is an individual-study appendix (ISA) under master protocol J2N-MC-JZNY, and represents participants from the completed originator study, clinical study LOXO-BTK-18001/J2N-OX-JZNA. Participants in the originator study will have the opportunity to continue their assigned study intervention or continue their follow-up visits by transitioning to this study. This study will evaluate the long-term safety and efficacy of pirtobrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Are currently enrolled and active in the originator study, LOXO-BTK-18001. A participant is considered active in the study if they are:

  * receiving study intervention
  * in the short-term follow-up period, or
  * in the long-term follow-up period

Exclusion Criteria:

* Were a participant in the Phase 1b cohort of Study LOXO-BTK-18001

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with a Grade ≥3 treatment-emergent adverse events (TEAEs) | Time from the Date of the First Dose of Study Intervention (Study Day 1) through 30 Days (+ 7-day window) After the Date of the Last Dose of Study Intervention or The First Date Starting a New Anticancer Therapy, whichever is Earlier

SECONDARY OUTCOMES:
Overall Survival | Time from Enrollment from the Originator Study until Death from Any Cause (Up to 93 Months)
  Overall survival is defined as the time from enrollment from the originator study until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- United States (17):
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - The Emory Clinic, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic- Minnesota, Rochester, Minnesota
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Cayuga Cancer Center, Ithaca, New York
  - Northwell Health, Lake Success, New York
  - Memorial Sloan-Kettering Cancer Center (MSKCC) - New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Flinders Medical Centre, Adelaide
  - Peter MacCallum Cancer Centre, Melbourne
  - Linear Clinical Research, Victoria
- CHU de Nantes - Hotel Dieu, Nantes, France
- Italy (2):
  - IRCCS-AOU di Bologna-Policlinico S.Orsola-Malpighi, Bologna
  - Ospedale San Raffaele, Milan
- Japan (6):
  - Nagoya Medical Center, Aichi-Ken
  - National Cancer Center Hospital, Cho-ku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Tokai University Hospital- Isehara Campus, Isehara
  - Tohoku University Hospital, Miyagi-Ken
  - Hokkaido University Hospital, Sapporo
- Poland (2):
  - Pratia MCM Krakow, Krakow
  - Instytut Hermatologii I Transfuzjologii, Warsaw
- Seoul National University Hospital, Seoul, South Korea
- United Kingdom (3):
  - St James's University Hospital, Leeds
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/